CLINICAL TRIAL: NCT00898508
Title: Blood Tumor Markers for Molecular Diagnosis of Breast Diseases and Monitoring of Breast Cancer Treatment and Follow-up
Brief Title: Studying Blood and Tumor Tissue Samples in Women With Invasive Breast Cancer, Ductal or Lobular Carcinoma in Situ, or Benign Breast Disease
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 04125; P30CA033572 (NIH); CHNMC-04125 (Registry Identifier: NCI PDQ); CDR0000628766 (Registry Identifier: NCI)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; invasive lobular breast carcinoma; ductal breast carcinoma in situ; lobular breast carcinoma in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Fluorescent Antibody Technique; Immunohistochemistry; Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample and biopsy tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal benign breast disease or ductal carcinoma in situ
  Interventions: Genetic: gene expression analysis; Genetic: mutation analysis; Genetic: proteomic profiling; Genetic: reverse transcriptase-polymerase chain reaction; Other: fluorescent antibody technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Other: medical chart review; Procedure: quality-of-life assessment
- Invasive breast cancer
  Interventions: Genetic: gene expression analysis; Genetic: mutation analysis; Genetic: proteomic profiling; Genetic: reverse transcriptase-polymerase chain reaction; Other: fluorescent antibody technique; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Other: medical chart review; Procedure: quality-of-life assessment

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: proteomic profiling
Genetic: reverse transcriptase-polymerase chain reaction
Other: fluorescent antibody technique
Other: immunohistochemistry staining method
  Groups: Normal benign breast disease or ductal carcinoma in situ
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry
Other: medical chart review
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Collecting and storing samples of blood and tumor tissue from patients with cancer to test in the laboratory may help the study of cancer in the future.

PURPOSE: This clinical trial is studying blood and tumor tissue samples in women with invasive breast cancer, ductal carcinoma in situ, lobular carcinoma in situ, or benign breast disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish a specimen bank from peripheral blood specimens collected from women with a full spectrum of breast disease (invasive breast cancer [IBC], ductal or lobular carcinoma in situ [CIS], or benign breast disease [BBD]) with standardized clinical follow up and serial specimen collection for those with IBC.
* To determine the ability of quantitative real-time reverse-transcriptase PCR (qRT-PCR) to discriminate between patients with IBC, CIS, and BBD by comparing baseline assay values from pre-biopsy specimens to the histologic diagnosis.
* To determine the ability of qRT-PCR to predict treatment response by comparing serial assay values from patients with evaluable IBC to their objective response.
* To determine the ability of qRT-PCR to predict relapse by comparing the serial assay values from all patients with IBC to their disease status.
* To determine the ability of qRT-PCR to perform as an independent prognostic factor by comparing baseline assay values from all patients with IBC to their disease status, stratified by known breast cancer prognostic factors.

Secondary

* To perform exploratory studies identifying potential targets for novel nucleic acid and proteomic-based early detection assays.

OUTLINE: Patients undergo baseline peripheral blood specimen collection pre-biopsy and then periodically for up to 10 years. Specimens are analyzed for circulating tumor cells via quantitative real-time reverse-transcriptase PCR, immunofluorescence, and bidirectional pyrophosphorolysis-activated polymerization allele-specific amplification; and for protein profiles via mass spectometry, liquid chromatography, enzyme digestion, and tandem mass spectometry. Patients' tumor tissue (invasive breast cancer [IBC] only) is analyzed for p53 via IHC. Medical records are reviewed periodically.

Patients with IBC complete a quality of life assessment at baseline and every 6 months for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-confirmed diagnosis of one of the following:

  * Stage I-IV infiltrating ductal or infiltrating lobular carcinoma

    * Patients with early-stage disease must not have started systemic treatment; if no systemic treatment is planned, patients must be either preoperative or ≤ 120 days since definitive breast surgery
    * Patients with locally advanced disease must be scheduled for neoadjuvant chemotherapy prior to initiation of systemic treatment
  * Ductal carcinoma in situ
  * Lobular carcinoma in situ
  * Benign breast disease

    * Proliferative or non-proliferative
    * With or without atypia

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Not pregnant
* No prior invasive cancer diagnosis within the past 5 years except for squamous cell or basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic therapy (chemotherapy or hormonal therapy) for patients with stage I-III disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: City of Hope New patients
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2005-08; Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Establishment of a specimen bank | 5 Years of specimen collection
Ability of the quantitative real-time reverse-transcriptase PCR (qRT-PCR) to distinguish between biopsy benign and malignant results | 5 years
Ability of the qRT-PCR to predict treatment response | 5 years
Ability of the qRT-PCR to predict relapse | 5 years
Ability of the qRT-PCR to perform as an independent prognostic factor | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hickey, Ph.D., Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California